CLINICAL TRIAL: NCT02230137
Title: Impact of Mobile Phone Short Text Messages on the Glycaemic Control of Adolescents With Poorly Controlled Type 1 Diabetes.
Brief Title: Text Message for Adolescents With Poorly Controlled Type 1 Diabetes
Acronym: Diabeto-SMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014-A00915-42
Record Dates: First submitted 2014-08-07; First posted 2014-09-03 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Type 1 Diabetes
Keywords: adolescents; type 1 diabetes; poorly controlled; SMS; Improve glycaemic control; HbA1c reduction; poorly controlled type 1 diabetic adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Text message arm (Experimental)
  Interventions: Behavioral: Text message arm
- No text message arm (No Intervention)

INTERVENTIONS:
Behavioral: Text message arm — Text message sent before each injection of insulin
  Other Names: Mobile phone short text message
  Arms: Text message arm

SUMMARY:
The purpose of this study is to assess HbA1c reduction after supportive care by SMS among adolescents with poorly controlled type 1 diabetes.

DETAILED DESCRIPTION:
In 2010, the number of children with type 1 diabetes in France is estimated at 12,000 with 60% of them aged 12 to 17 years. Compliance is a major issue during adolescence. Mobile text message is one of the strategies to enhance adherence. The main aim of this study is to assess HbA1c reduction after a 6 month SMS support among adolescents with poorly controlled type 1 diabetes. Adherence and quality of life will also be assessed at the end of the trial. This study is a prospective randomized monocentric trial. Sixty adolescents with type 1 diabetes and HbA1c equal or higher than 8.5 % will be randomized according to the method of Zelen in two groups : standard treatment versus standard treatment plus support by SMS. The patients will receive one SMS before each injection of insulin.

ELIGIBILITY:
Inclusion Criteria:

* aged between 12 and 21 years old
* with type 1 diabetes for more than 6 months
* HbA1c at enrollment > 8.5%
* non-opposition of one of the parents
* previous medical exam (art. L.1121-11 du CSP)
* Possible follow-up for 6 months
* social welfare coverage
* Adolescents with a mobile phone, able to receive short text message

Exclusion Criteria:

* aged less than 12 or higher than 21 years old
* with HbA1c at enrollment < 8.5%
* pregnancy
* psychiatric disease
* do not understand french

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2015-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
HbA1c level | 6 months

SECONDARY OUTCOMES:
HbA1c level | 3 months
Compliance | 3 months
  blood glucose level
Compliance | 6 months
  blood glucose level
Quality of life | 3 months
  PedsQL version 4.0
Quality of life | 6 months
  PedsQL version 4.0
Satisfaction survey | 6 months
  7 items for patients randomized in the "Text message arm"

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Tréluyer, MD, PhD, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP Necker, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Louch G, Dalkin S, Bodansky J, Conner M. An exploratory randomised controlled trial using short messaging service to facilitate insulin administration in young adults with type 1 diabetes. Psychol Health Med. 2013;18(2):166-74. doi: 10.1080/13548506.2012.689841. Epub 2012 May 30. PMID 22646659
- [Background] Benhamou PY, Melki V, Boizel R, Perreal F, Quesada JL, Bessieres-Lacombe S, Bosson JL, Halimi S, Hanaire H. One-year efficacy and safety of Web-based follow-up using cellular phone in type 1 diabetic patients under insulin pump therapy: the PumpNet study. Diabetes Metab. 2007 Jun;33(3):220-6. doi: 10.1016/j.diabet.2007.01.002. Epub 2007 Mar 28. PMID 17395516
- [Background] Rami B, Popow C, Horn W, Waldhoer T, Schober E. Telemedical support to improve glycemic control in adolescents with type 1 diabetes mellitus. Eur J Pediatr. 2006 Oct;165(10):701-5. doi: 10.1007/s00431-006-0156-6. Epub 2006 May 3. PMID 16670859
- [Derived] Ibrahim N, Treluyer JM, Briand N, Godot C, Polak M, Beltrand J. Text message reminders for adolescents with poorly controlled type 1 diabetes: A randomized controlled trial. PLoS One. 2021 Mar 15;16(3):e0248549. doi: 10.1371/journal.pone.0248549. eCollection 2021. PMID 33720997